CLINICAL TRIAL: NCT06970236
Title: Impact of an In-hospital Exercise Program on the Health of Patients With Ocular Melanoma Undergoing Plaque Brachytherapy: A Randomized Controlled Trial
Brief Title: Resistance Exercise in Patients With Ocular Melanoma
Acronym: IHOPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Joaquín Calatayud Villalba, Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IHOPE-2025
Record Dates: First submitted 2025-03-27; First posted 2025-05-14 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Ocular Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention Group (Experimental): Participants on this group will follow the exercise intervention mentioned in the protocol.
  Interventions: Other: Exercise
- Control Group (No Intervention): Patients in the control group will follow the hospital's conventional protocol during the hospitalization days, which consists in isolated bed rest.

INTERVENTIONS:
Other: Exercise — Daily session during hospitalization. To carry out the training session, elastic bands (TheraBand CLX Consecutive Loops; TheraBand, Akron, OH) with resistance graded from very low to very high (i.e, yellow, red, green, blue, black, silver and gold) will be used. On each day, each exercise will start with 3 sets of two repetitions as a warm-up and to calculate the appropriate intensity. The intensity will be that at which the patient reports a perceived exertion of 5-6 of 10 at the Borg CR10 scale after two repetitions. For each exercise, one set will be completed until task failure is achieved.If in any of the exercises the patient perceives this intensity only with the weight of his own limb or body weight, the exercise will be performed without elastic bands.
  Arms: Exercise Intervention Group

SUMMARY:
Choroidal melanoma (CM) is one of the most common intraocular cancers worldwide. During treatment with episcleral brachytherapy, patients require a week of hospitalization in isolation. The primary aim of this study will be to investigate the effects of resistance training during hospitalization on health-related blood biomarkers in CM patients. Our secondary aim will be to assess changes in physical function tests, quality of life and anxiety and depression. Candidates for this study will be patients undergoing CM treatment at the "Hospital Universitari i Politècnic La Fe" of Valencia.

DETAILED DESCRIPTION:
Candidates of the present study will be adults with CM diagnose and treated with plaque brachytherapy undergoing in "Hospital Universitari i Politècnic La Fe" (Valencia). All the participants will be informed about the objectives and content of the investigation and written informed consent will be obtained. Participants will be excluded if they (1) present a health status that forbids high intensity resistance training, (2) have any unsteady cardiac illness, (3) have serious metabolic disorder or if (4) they have any important orthopaedic disorder impeding exercise. The study will conform to the Declaration of Helsinki and will be approved by the Ethical Committee of "Hospital Universitari i Politècnic de La Fe".

A randomized controlled trial with two parallel groups is planned: a control group following the hospital's standard protocol (usual care) and an intervention group in which patients will complete a daily resistance training session during hospitalization. During the 5-7 days of treatment, where participants are going to be isolated in a room without human contact, are going to perform a daily session of exercise during about 30 minutes. The exercises will be supervised by a trained physician. To carry out the training session, elastic resistance bands will be used. On each day, each exercise will start with 3 sets of two repetitions as a warm-up and to calculate the appropriate intensity. The intensity will be that at which the patient reports a perceived exertion of 5-6 of 10 at the Borg CR10 scale after two repetitions. For each exercise, one set will be completed until task failure is achieved.If in any of the exercises the patient perceives this intensity only with the weight of his own limb or body weight, the exercise will be performed without elastic bands.

To observe the effects of the intervention, various blood tests, functional, quality-of-life and anxiety and depression assessments will be conducted before and after the program, as well as one-month post-hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Adults with Choroidal Melanoma diagnose and treated with plaque brachytherapy undergoing in "Hospital Universitari i Politècnic La Fe" (Valencia).

Exclusion Criteria:

* Present a health status that forbids high intensity resistance training.
* Have any unsteady cardiac illness.
* Have serious metabolic disorder.
* Have any important orthopaedic disorder impeding exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Blood biomarkers: glucose | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in milligrams/deciliter (mg/dl).
Blood biomarkers: urea | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in milligrams/deciliter (mg/dl).
Blood biomarkers: creatinine | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in milligrams/deciliter (mg/dl).
Blood biomarkers: glomerular filtration | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in milliliters/minutes/1,73 (ml/min/1,73).
Blood biomarkers: total bilirubin | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in milligrams/deciliter (mg/dl).
Blood biomarkers: aspartate aminotransferase | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in units/liter (U/L).
Blood biomarkers: alanine aminotransferase | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in units/liter (U/L).
Blood biomarkers: alkaline phosphatase | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in units/liter (U/L).
Blood biomarkers: lactate dehydrogenase | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in units/liter (U/L).
Blood biomarkers: creatine kinase | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in units/liter (U/L).
Blood biomarkers: total proteins | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in grams/deciliter (g/dl).
Blood biomarkers: albumin | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in grams/deciliter (g/dl).
Blood biomarkers: C-reactive protein | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Inflammatory response marker measured in milligrams/liter (mg/L).
Blood biomarkers: interleukin 6 | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Inflammatory response marker measured in picograms/milliliter (pg/ml).
Blood biomarkers: calcium | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in milligrams/deciliter (mg/dl).
Blood biomarkers: albumine-corrected calcium | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in milligrams/deciliter (mg/dl).
Blood biomarkers: chloride | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in milliequivalents/liter (mEq/L).
Blood biomarkers: sodium | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in milliequivalents/liter (mEq/L).
Blood biomarkers: potassium | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in milliequivalents/liter (mEq/L).
Blood biomarkers: total cholesterol | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in milligrams/deciliter (mg/dl).
Blood biomarkers: HDL cholesterol | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in milligrams/deciliter (mg/dl).
Blood biomarkers: LDL cholesterol | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in milligrams/deciliter (mg/dl).
Blood biomarkers: no HDL cholesterol | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in milligrams/deciliter (mg/dl).
Blood biomarkers: triglycerides | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in milligrams/deciliter (mg/dl).
Blood biomarkers: hematies | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in x10^6/microliter (x10^6/µL).
Blood biomarkers: hemoglobin | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in grams/deciliter (g/dl).
Blood biomarkers: hematocrit | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in percentage (%).
Blood biomarkers: mean corpuscular volume | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in femtoliters (fL).
Blood biomarkers: mean corpuscular hemoglobine | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in picograms (pg).
Blood biomarkers: mean corpuscular hemoglobin concentration | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in grams/deciliter (g/dl).
Blood biomarkers: red cell distribution width - standard deviation | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in femtoliters (fL).
Blood biomarkers: red cell distribution width - coefficient of variation | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in percentage (%).
Blood biomarkers: erythroblasts | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in percentage (%).
Blood biomarkers: leukocytes | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in x10^3/microliter (x10^3/µL).
Blood biomarkers: neutrophils | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in x10^3/microliter (x10^3/µL).
Blood biomarkers: lymphocytes | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in x10^3/microliter (x10^3/µL).
Blood biomarkers: monocytes | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in x10^3/microliter (x10^3/µL).
Blood biomarkers: eosinophils | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in x10^3/microliter (x10^3/µL).
Blood biomarkers: basophils | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in x10^3/microliter (x10^3/µL).
Blood biomarkers: neutrophils % | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in percentage (%).
Blood biomarkers: lymphocytes % | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in percentage (%).
Blood biomarkers: monocytes % | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in percentage (%).
Blood biomarkers: eosinophils % | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in percentage (%).
Blood biomarkers: basophils % | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in percentage (%).
Blood biomarkers: immature granulocytes % | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in percentage (%).
Blood biomarkers: platelets | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in x10^3/microliter (x10^3/µL).
Blood biomarkers: mean platelet volume | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in femtoliters (fL).
Blood biomarkers: platelet distribution width | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in femtoliters (fL).
Blood biomarkers: platelet large cell ratio | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in percentage (%).
Blood biomarkers: prothrombin time | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in seconds (sec).
Blood biomarkers: prothrombin time ratio | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker.
Blood biomarkers: Quick index | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in percentage (%).
Blood biomarkers: activated partial thromboplastin time | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in seconds (sec).
Blood biomarkers: activated partial thromboplastin time ratio | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker.
Blood biomarkers: derived fibrinogen | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Blood marker measured in milligrams/deciliter (mg/dl).
Blood biomarkers: procalcitonin | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Inflammatory response markers measured in nanograms/milliliter (ng/ml).
Blood biomarkers: glycated hemoblobin A1c | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in percentage (%).
Blood biomarkers: estimated average glucose | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Metabolic and lipidic response marker measured in milligrams/deciliter (mg/dl).
Blood biomarkers: carcinoembryonic antigen | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Tumor marker measured in nanograms per milliliter (ng/ml).
Blood biomarkers: S-100 | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  Tumor markers measured in micrograms per liter (µg/L).

SECONDARY OUTCOMES:
EORTC_C30 | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  The patient self-reported outcomes comprised the EORTC_ C30 questionnaire. This survey assesses various dimensions of quality of life.
EORTC_OPT30 | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  The patient self-reported outcomes comprised also the complementary EORTC_ OPT30 module specifically designed for patients with eye cancer. This survey assesses various dimensions of quality of life, and the OPT30 module has a particular focus on evaluating visual functioning limitations.
HADS questionnaire | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  The Hospital Anxiety and Depression Scale (HADS) will be used to measure symptoms of anxiety (HADS Anxiety) and depression (HADS Depression).
Physical activity levels | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  The patients will be also asked about their levels of physical activity prior to hospitalization (minutes/week during the last month).
TUG test | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  To evaluate agility/coordination, the timed-up-and-go-test (TUG) will be used to, which consists of rising from a chair on command, walking a distance of 3 m, turning around, and walking back to the chair as fast as possible.
30s StS Test | At baseline, during hospital discharge day (5-7 days after baseline measure) and one month after hospital discharge.
  To assess muscle strength of lower limbs (endurance strength), the patient will be performed the 30-s sit-to-stand test (30 s StS), which is to stand up and sit down as many times as possible in 30 s.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari i Politècnic de La Fe, Valencia, Spain, Spain

IPD SHARING:
Plan to Share IPD: No